CLINICAL TRIAL: NCT01170455
Title: Nasal Intubation Using the Blind Intubation Device:a Prospective,Randomized,Controlled Comparison With the Direct Laryngoscope
Brief Title: Nasal Intubation Using the Blind Intubation Device
Acronym: BID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Shanghai Ninth People's Hospital, Hong Jiang
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shanghai 9th People's Hospital
Record Dates: First submitted 2010-07-21; First posted 2010-07-27 (Estimated); Last update posted 2010-10-29 (Estimated); Status verified 2010-09

CONDITIONS: Intubation
Keywords: nasal; intubation; direct laryngoscope; blind; normal airway

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blind Intubation Device (Experimental)
  Interventions: Device: Blind Intubation Device
- Direct laryngoscope (Active Comparator)
  Interventions: Device: Macintosh laryngoscope

INTERVENTIONS:
Device: Macintosh laryngoscope — nasal intubation with macintosh laryngoscope after general anesthesia induction
  Arms: Direct laryngoscope
Device: Blind Intubation Device — nasal intubation using Blind Intubation Device after general anesthesia induction
  Arms: Blind Intubation Device

SUMMARY:
The purpose of this study is to determine whether nasal tracheal intubation using Blind Intubation Device is safe and effective in anesthetized patients with Mallampati class 3

DETAILED DESCRIPTION:
The Blind Intubation Device (BID,Anhui Xiao Shan Hygienic Material Co.Ltd,Jixi County,China) is newly introduced for awake nasal intubation using a transillumination principle. For oral and maxillofacial surgery patients with anticipated difficult airways, the BID has a high rate of successful awake nasal intubation.Since the BID is more readily accessible,disposable and considerably less expensive,these advantages speak well for its use in China.However,to date,there is no study on its usage in anesthetized patients.The investigators hypothesized that a BID would be effective for nasal intubation in anesthetized patients with high Mallampati class and would result in fewer hemodynamic responses. To examine our hypothesis, the investigators would like to perform a prospective,randomized,controlled study to compare the effectiveness of the BID technique with a direct laryngoscope for nasal intubation in anesthetized patients with Mallampati class 3. The primary outcome measures are the hemodynamic changes during intubation. The investigators also would like to compare the intubation time required and associated airway complications in both groups as our second outcome.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1-2
* Scheduled for oral and maxillofacial surgery under general anesthesia with nasotracheal intubation
* mallampati score 3

Exclusion Criteria:

* ASA physical status 3-4
* Patients with a history of intraoral,upper airway and neck surgeries
* Patients with a history of chronic respiratory, cardiovascular or any other systemic diseases
* morbid obesity
* neck scars
* mallampati score 4,inter-incisor distance<3cm, thyromental distance<6cm
* unstable cervical spine
* relevant drug allergy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Hemodynamic changes | 1 min before general anesthesia induction
Hemodynamic changes | 5 min after general anesthesia induction
Hemodynamic changes | 30s from nasal intubation start
Hemodynamic changes | 1 min after nasal intubation
Hemodynamic changes | 2 min after nasal intubation
Hemodynamic changes | 3 min after nasal intubation
hemodynamic changes | 4 min from nasal intubation start
hemodynamic changes | 5 min from nasal intubation start

SECONDARY OUTCOMES:
intubation time required | 0 min after nasal intubation
  from taking of the intubation device to successful intubation
immediate associated airway complications | 5 min after nasal intubation
  mucosal injury,dental injury,airway injury,bleeding, etc
24h associated airway complications | 24h after intubation
  sore throat, hoarseness, etc

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Hong, PhD,MD, Study Chair — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University; Sun Yu, PhD,MD, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University; Liu J Xing, MD, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University; Xu Hui, MD, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University; Huang Yan, MD, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University; Zhu Y Sen, MD, Study Director — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Department of Anesthesiology, Shanghai 9th People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Sun Y, Liu JX, Jiang H, Zhu YS, Xu H, Huang Y. Cardiovascular responses and airway complications following awake nasal intubation with blind intubation device and fibreoptic bronchoscope: a randomized controlled study. Eur J Anaesthesiol. 2010 May;27(5):461-7. doi: 10.1097/EJA.0b013e328332845a. PMID 20090540
- [Background] Sun Y, Jiang H, Zhu Y, Xu H, Huang Y. Blind intubation device for nasotracheal intubation in 100 oral and maxillofacial surgery patients with anticipated difficult airways: a prospective evaluation. Eur J Anaesthesiol. 2009 Sep;26(9):746-51. doi: 10.1097/EJA.0b013e32832b13a2. PMID 19451824
- [Derived] Sun Y, Liu JX, Zhu YS, Xu H, Huang Y, Jiang H. Nasotracheal intubation using the Blind Intubation Device in anaesthetised adults with Mallampati class 3: a comparison with the Macintosh laryngoscope. Eur J Anaesthesiol. 2011 Nov;28(11):774-80. doi: 10.1097/EJA.0b013e328349a9f9. PMID 21885980